CLINICAL TRIAL: NCT04406389
Title: InterMediate ProphylACtic Versus Therapeutic Dose Anticoagulation in Critically Ill Patients With COVID-19: A Prospective Randomized Study (The IMPACT Trial)
Brief Title: Anticoagulation in Critically Ill Patients With COVID-19 (The IMPACT Trial)
Acronym: IMPACT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-04021936
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: COVID-19; Anticoagulation
MeSH Terms: conditions — COVID-19 | interventions — enoxaparin sodium; Enoxaparin; Heparin; Fondaparinux; argatroban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermediate Dose Prophylaxis (Active Comparator): Subjects will receive one of the following interventions, at their physician's discretion:
  * Enoxaparin 0.5 mg/kg subcutaneously every 12 hours if creatinine clearance greater than or equal to 30 ml/min
  * Enoxaparin 0.5 mg/kg subcutaneously every 24 hours if creatinine clearance less than 30 mL/min
  * If patient develops acute kidney injury: unfractionated heparin 7,500 units subcutaneously every 8 hours.
  * Fondaparinux (if history of heparin-inducted thrombocytopenia [HIT]) 2.5 mg daily subcutaneously
  Interventions: Drug: Enoxaparin sodium; Drug: Unfractionated heparin; Drug: Fondapariniux
- Therapeutic Dose Anticoagulation (Experimental): Subjects will receive one of the following interventions, at their physician's discretion:
  * Unfractionated heparin (UFH) to target anti-Xa level 0.3 -0.7 IU/mL or activated partial thromboplastin time (aPTT) (according to institutional protocol).
  * Enoxaparin 1 mg/kg subcutaneously every 12 hours
  * Argatroban (if heparin-induced thrombocytopenia [HIT]), dosed according to institutional protocol.
  * Fondaparinux (if HIT and creatinine clearance greater than or equal to 50 ml/min) dosed by weight:
    * ≥100 kg: 10 mg daily
    * <100 kg but ≥50 kg: 7.5 mg daily
    * <50 kg: 5 mg daily
  Interventions: Drug: Enoxaparin sodium; Drug: Unfractionated heparin; Drug: Fondapariniux; Drug: Argatroban

INTERVENTIONS:
Drug: Enoxaparin sodium — Intermediate Dose Prophylaxis Arm:
  0.5 mg/kg subcutaneously every 12 hours if creatinine clearance greater than or equal to 30 ml/min --OR-- 0.5 mg/kg subcutaneously every 24 hours if creatinine clearance less than 30 ml/min
  Therapeutic Dose Anticoagulation Arm:
  1 mg/kg subcutaneously every 12 hours
  Other Names: Lovenox
Drug: Unfractionated heparin — Intermediate Dose Prophylaxis Arm:
  7,500 units subcutaneously every 8 hours
  Therapeutic Dose Anticoagulation Arm:
  Dosed to target anti-Xa level 0.3 - 0.7 IU/mL or activated partial thromboplastin time (aPTT), according to institutional protocol
  Other Names: Sodium heparin
Drug: Fondapariniux — Intermediate Dose Prophylaxis Arm:
  2.5 mg daily subcutaneously
  Therapeutic Dose Anticoagulation Arm:
  Dose by weight:
  * If greater than or equal to 100 kg: 10 mg daily
  * If less than 100 kg but greater than or equal to 50 kg: 7.5 mg daily
  * If less than 50 kg: 5 mg daily
  Other Names: Arixtra
Drug: Argatroban — Therapeutic Dose Anticoagulation Arm:
  Dosed according to institutional protocol
  Arms: Therapeutic Dose Anticoagulation

SUMMARY:
The purpose of this study is to determine if therapeutic dose anticoagulation (experimental group) improves 30-day mortality in participants with COVID-19 compared to those patients receiving the intermediate dose prophylaxis (control group). Following screening, subjects will be randomized 1:1 to intermediate dose prophylaxis or therapeutic dose anticoagulation treatment arms.Treatment will continue for 28 days, followed by a 6 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* COVID-19 positive on (RT-PCR) nasopharyngeal swab, or suspected COVID-19 infection with detectable SARS-CoV-2 IgG or IgM.
* Intensive care unit (ICU) patient or non-ICU patient on invasive mechanical ventilation, BiPAP, 100% non-rebreather mask, or high flow oxygen or supplemental oxygen of at least 4 liters per minute nasal cannula.
* D dimer level greater than 700 ng/mL (3 times the upper limit of normal).

Exclusion Criteria:

* Objectively documented deep vein thrombosis or pulmonary embolism
* Patients in whom there is very high suspicion for pulmonary embolism and are on full-dose anticoagulation as per the treating physician
* Platelets <30,000 not due to disseminated intravascular coagulation (DIC), based on the International Society of Thrombosis and Haemostasis (ISTH) criteria and American Society of Hematology (ASH) Frequently Asked Questions
* Active bleeding that poses a contraindication to therapeutic anticoagulation in the opinion of the investigator.
* History of bleeding diathesis (e.g., hemophilia, severe von Willebrand disease, severe thrombocytopathy)
* History of intracranial hemorrhage in the last 90 days
* History of ischemic stroke in the past 2 weeks
* Major neurosurgical procedure in the past 30 days
* Cardiothoracic surgery in the past 30 days
* Intra-abdominal surgery in the past 30 days
* Intracranial malignancy
* Patients who require therapeutic anticoagulation for other reasons like atrial fibrillation, deep venous thrombosis, pulmonary embolism, or antiphospholipid syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria T DeSancho, MD, MSc, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang N, Li D, Wang X, Sun Z. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 Apr;18(4):844-847. doi: 10.1111/jth.14768. Epub 2020 Mar 13. PMID 32073213
- [Background] Tang N, Bai H, Chen X, Gong J, Li D, Sun Z. Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy. J Thromb Haemost. 2020 May;18(5):1094-1099. doi: 10.1111/jth.14817. Epub 2020 Apr 27. PMID 32220112
- [Background] Xiong TY, Redwood S, Prendergast B, Chen M. Coronaviruses and the cardiovascular system: acute and long-term implications. Eur Heart J. 2020 May 14;41(19):1798-1800. doi: 10.1093/eurheartj/ehaa231. No abstract available. PMID 32186331
- [Background] Young E. The anti-inflammatory effects of heparin and related compounds. Thromb Res. 2008;122(6):743-52. doi: 10.1016/j.thromres.2006.10.026. Epub 2007 Aug 28. PMID 17727922
- [Background] Esmon CT. Targeting factor Xa and thrombin: impact on coagulation and beyond. Thromb Haemost. 2014 Apr 1;111(4):625-33. doi: 10.1160/TH13-09-0730. Epub 2013 Dec 12. PMID 24336942
- [Background] Poterucha TJ, Libby P, Goldhaber SZ. More than an anticoagulant: Do heparins have direct anti-inflammatory effects? Thromb Haemost. 2017 Feb 28;117(3):437-444. doi: 10.1160/TH16-08-0620. Epub 2016 Dec 15. PMID 27975101
- [Background] Hanify JM, Dupree LH, Johnson DW, Ferreira JA. Failure of chemical thromboprophylaxis in critically ill medical and surgical patients with sepsis. J Crit Care. 2017 Feb;37:206-210. doi: 10.1016/j.jcrc.2016.10.002. Epub 2016 Oct 11. PMID 27969572
- [Background] Thachil J. The versatile heparin in COVID-19. J Thromb Haemost. 2020 May;18(5):1020-1022. doi: 10.1111/jth.14821. Epub 2020 Apr 27. No abstract available. PMID 32239799
- [Background] Cui S, Chen S, Li X, Liu S, Wang F. Prevalence of venous thromboembolism in patients with severe novel coronavirus pneumonia. J Thromb Haemost. 2020 Jun;18(6):1421-1424. doi: 10.1111/jth.14830. Epub 2020 May 6. PMID 32271988
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Helms J, Tacquard C, Severac F, Leonard-Lorant I, Ohana M, Delabranche X, Merdji H, Clere-Jehl R, Schenck M, Fagot Gandet F, Fafi-Kremer S, Castelain V, Schneider F, Grunebaum L, Angles-Cano E, Sattler L, Mertes PM, Meziani F; CRICS TRIGGERSEP Group (Clinical Research in Intensive Care and Sepsis Trial Group for Global Evaluation and Research in Sepsis). High risk of thrombosis in patients with severe SARS-CoV-2 infection: a multicenter prospective cohort study. Intensive Care Med. 2020 Jun;46(6):1089-1098. doi: 10.1007/s00134-020-06062-x. Epub 2020 May 4. PMID 32367170
- [Background] Middeldorp S, Coppens M, van Haaps TF, Foppen M, Vlaar AP, Muller MCA, Bouman CCS, Beenen LFM, Kootte RS, Heijmans J, Smits LP, Bonta PI, van Es N. Incidence of venous thromboembolism in hospitalized patients with COVID-19. J Thromb Haemost. 2020 Aug;18(8):1995-2002. doi: 10.1111/jth.14888. Epub 2020 Jul 27. PMID 32369666
- [Background] Goyal P, Choi JJ, Pinheiro LC, Schenck EJ, Chen R, Jabri A, Satlin MJ, Campion TR Jr, Nahid M, Ringel JB, Hoffman KL, Alshak MN, Li HA, Wehmeyer GT, Rajan M, Reshetnyak E, Hupert N, Horn EM, Martinez FJ, Gulick RM, Safford MM. Clinical Characteristics of Covid-19 in New York City. N Engl J Med. 2020 Jun 11;382(24):2372-2374. doi: 10.1056/NEJMc2010419. Epub 2020 Apr 17. No abstract available. PMID 32302078
- [Background] Paranjpe I, Fuster V, Lala A, Russak AJ, Glicksberg BS, Levin MA, Charney AW, Narula J, Fayad ZA, Bagiella E, Zhao S, Nadkarni GN. Association of Treatment Dose Anticoagulation With In-Hospital Survival Among Hospitalized Patients With COVID-19. J Am Coll Cardiol. 2020 Jul 7;76(1):122-124. doi: 10.1016/j.jacc.2020.05.001. Epub 2020 May 6. No abstract available. PMID 32387623
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 subject signed consent but failed screening and was not randomized.
Groups:
- Intermediate Dose Prophylaxis: Subjects will receive one of the following interventions, at their physician's discretion:
  * Enoxaparin 0.5 mg/kg subcutaneously every 12 hours if creatinine clearance greater than or equal to 30 ml/min
  * Enoxaparin 0.5 mg/kg subcutaneously every 24 hours if creatinine clearance less than 30 mL/min
  * If patient develops acute kidney injury: unfractionated heparin 7,500 units subcutaneously every 8 hours.
  * Fondaparinux (if history of heparin-inducted thrombocytopenia [HIT]) 2.5 mg daily subcutaneously
  Enoxaparin sodium: Intermediate Dose Prophylaxis Arm:
  0.5 mg/kg subcutaneously every 12 hours if creatinine clearance greater than or equal to 30 ml/min --OR-- 0.5 mg/kg subcutaneously every 24 hours if creatinine clearance less than 30 ml/min
  Therapeutic Dose Anticoagulation Arm:
  1 mg/kg subcutaneously every 12 hours
  Unfractionated heparin: Intermediate Dose Prophylaxis Arm:
  7,500 units subcutaneously every 8 hours
  Therapeutic Dose Anticoagulation Arm:
  Dosed to target anti-Xa level 0.3 - 0.7 IU/mL or activated partial thromboplastin time (aPTT), according to institutional protocol
  Fondapariniux: Intermediate Dose Prophylaxis Arm:
  2.5 mg daily subcutaneously
  Therapeutic Dose Anticoagulation Arm:
  Dose by weight:
  * If greater than or equal to 100 kg: 10 mg daily
  * If less than 100 kg but greater than or equal to 50 kg: 7.5 mg daily
  * If less than 50 kg: 5 mg daily
- Therapeutic Dose Anticoagulation: Subjects will receive one of the following interventions, at their physician's discretion:
  * Unfractionated heparin (UFH) to target anti-Xa level 0.3 -0.7 IU/mL or activated partial thromboplastin time (aPTT) (according to institutional protocol).
  * Enoxaparin 1 mg/kg subcutaneously every 12 hours
  * Argatroban (if heparin-induced thrombocytopenia [HIT]), dosed according to institutional protocol.
  * Fondaparinux (if HIT and creatinine clearance greater than or equal to 50 ml/min) dosed by weight:
    * 100kg: 10 mg daily <100kg but ≥50 kg: 7.5 mg daily <50kg: 5 mg daily
  Enoxaparin sodium: Intermediate Dose Prophylaxis Arm:
  0.5 mg/kg subcutaneously every 12 hours if creatinine clearance greater than or equal to 30 ml/min, OR 0.5 mg/kg subcutaneously every 24 hours if creatinine clearance less than 30 ml/min
  Therapeutic Dose Anticoagulation Arm:
  1 mg/kg subcutaneously every 12 hours
  Unfractionated heparin: Intermediate Dose Prophylaxis Arm:
  7,500 units subcutaneously every 8 hours
  Therapeutic Dose Anticoagulation Arm:
  Dosed to target anti-Xa level 0.3 - 0.7 IU/mL or activated partial thromboplastin time (aPTT), according to institutional protocol
  Fondapariniux: Intermediate Dose Prophylaxis Arm:
  2.5mg daily subcutaneously
  Therapeutic Dose Anticoagulation Arm:
  Dose by weight:
  ≥100kg: 10 mg daily <100kg but ≥50 kg: 7.5 mg daily <50kg: 5 mg daily
  Argatroban: Therapeutic Dose Anticoagulation Arm:
  Dosed according to institutional protocol
Period: Overall Study
Arm/Group | Intermediate Dose Prophylaxis | Therapeutic Dose Anticoagulation
Started | 4 | 10
Completed | 4 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermediate Dose Prophylaxis | Therapeutic Dose Anticoagulation | Total
Number analyzed (Participants) | 4 | 10 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 7 | 8
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 14
Subject Location at Time of Randomization [Count of Participants; unit: Participants]
  Intensive Care Unit | 2 | 6 | 8
  Ward | 2 | 4 | 6
Respiratory Support at Time of Randomization [Count of Participants; unit: Participants]
  High Flow Nasal Cannula or Non-Invasive Ventilation (>15 L/min) | 1 | 6 | 7
  Invasive Mechanical Ventilation or ECMO | 1 | 2 | 3
  Supplemental Oxygen (<15L/min) | 2 | 2 | 4
Vasopressor Support at Time of Randomization [Count of Participants; unit: Participants]
  Subjects on Vasopressor Support | 0 | 2 | 2
  Subjects not on Vasopressor Support | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: 30-day Mortality
Description: Comparison of number of COVID-19 positive patients who have died within 30 days of starting treatment on each treatment arm
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Dose Prophylaxis | Therapeutic Dose Anticoagulation
Number analyzed (Participants) | 4 | 10
Participants | 0 | 2

2. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay in Days
Description: Comparison of length of ICU stay in days between each treatment arm.
Time Frame: 6 months
Population: This outcome measure is only assessing participants that had an ICU stay while participating in the study. Participants that never had an ICU stay are excluded from the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Intermediate Dose Prophylaxis | Therapeutic Dose Anticoagulation
Number analyzed (Participants) | 2 | 6
Days | 25.5 [10 to 41] | 25 [15 to 111]

3. Secondary Outcome: Number of Documented Venous Thromboembolism (VTE), Arterial Thrombosis (Stroke, Myocardial Infarction, Other) and Microthrombosis Events
Description: Comparison of number of documented VTE, arterial thrombosis and microthrombosis events on each treatment arm
Time Frame: 6 months
Measure: Number; unit: Count of Events
Arm/Group | Intermediate Dose Prophylaxis | Therapeutic Dose Anticoagulation
Number analyzed (Participants) | 4 | 10
Count of Events
  Venous Thromboembolism Events | 1 | 0
  Arterial Thrombosis Events | 1 | 0
  Microthrombosis Events | 0 | 1

4. Secondary Outcome: Number of Major and Clinically Relevant Non-major Bleeding Events
Description: Comparison of major and clinically-relevant non-major bleeding events on each treatment arm, as defined by the International Society of Thrombosis and Haemostasis (ISTH) criteria.
Time Frame: 6 months
Measure: Number; unit: Count of Events
Arm/Group | Intermediate Dose Prophylaxis | Therapeutic Dose Anticoagulation
Number analyzed (Participants) | 4 | 10
Count of Events
  Major Bleeding Events | 1 | 1
  Clinically Relevant Non-Major Bleeding Events | 1 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Description: Only adverse events (AEs) meeting the following criteria will be collected and reported:
  1. AEs related to bleeding (any major or clinically significant non-major bleeding) or thrombotic events (DVT/PE, stroke, myocardial infarction, peripheral embolism, skin thrombosis).
  2. Any AE that results in interruption or discontinuation of the assigned anticoagulant treatment.
  3. Any AE that meets the criteria for serious
Arm/Group | Intermediate Dose Prophylaxis | Therapeutic Dose Anticoagulation
All-Cause Mortality (participants affected / at risk) | 0/4 | 4/10
Serious Adverse Events (participants affected / at risk) | 1/4 | 4/10
Other Adverse Events (participants affected / at risk) | 1/4 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermediate Dose Prophylaxis (N=4) | Therapeutic Dose Anticoagulation (N=10)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic Event - Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
Multi-organ Failure (General disorders) | 0 (0) | 2 (2)
Gluteal Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Ischemic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermediate Dose Prophylaxis (N=4) | Therapeutic Dose Anticoagulation (N=10)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2)
Tracheostomy Site Bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders, Other - Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Navigational Note: - Respiratory, thoracic and mediastinal disorders - Other - Oropharyngeal bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The statistical analysis plan (and associated statistical power) was based on an expected sample size of 186 participants. As only 14 participants enrolled, this reduced sample size is not sufficient for the statistical analysis plan as written, and, therefore, only descriptive statistics are presented for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT04406389/Prot_SAP_000.pdf